CLINICAL TRIAL: NCT05052970
Title: A Phase Ⅰ Clinical Study of Mitoxantrone Hydrochloride Liposome Injection in Combination With Bortezomib and Dexamethasone in Patients With Relapsed or Refractory Multiple Myeloma
Brief Title: Mitoxantrone Hydrochloride Liposome Injection, Bortezomib and Dexamethasone in the Treatment of R/R MM
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: CSPC Zhongnuo Pharmaceutical (Shijiazhuang) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HE071-CSP-023
Record Dates: First submitted 2021-09-13; First posted 2021-09-22 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Relapsed or Refractory Multiple Myeloma
MeSH Terms: conditions — Recurrence; Multiple Myeloma | interventions — Bortezomib; Injections; dexamethasone acetate; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 12 mg/m ^ 2 dose group (ArmA) (Experimental): Patients with relapsed or refractory multiple myeloma will receive mitoxantrone hydrochloride liposome in combination with bortezomib and dexamethasone for 8 cycles (planned) (28 days per cycle). The dose of mitoxantrone hydrochloride liposome is 12 mg/m^2
  Interventions: Drug: Mitoxantrone Hydrochloride Liposome injection; Drug: Bortezomib for Injection; Drug: Dexamethasone Acetate Tablets
- 16 mg/m ^ 2 dose group (ArmB) (Experimental): Patients with relapsed or refractory multiple myeloma will receive mitoxantrone hydrochloride liposome in combination with bortezomib and dexamethasone for 8 cycles (planned) (28 days per cycle). The dose of mitoxantrone hydrochloride liposome is 16 mg/m^2
  Interventions: Drug: Mitoxantrone Hydrochloride Liposome injection; Drug: Bortezomib for Injection; Drug: Dexamethasone Acetate Tablets
- 20 mg/m ^ 2 dose group (ArmC) (Experimental): Patients with relapsed or refractory multiple myeloma will receive mitoxantrone hydrochloride liposome in combination with bortezomib and dexamethasone for 8 cycles (planned) (28 days per cycle). The dose of mitoxantrone hydrochloride liposome is 20 mg/m^2
  Interventions: Drug: Mitoxantrone Hydrochloride Liposome injection; Drug: Bortezomib for Injection; Drug: Dexamethasone Acetate Tablets

INTERVENTIONS:
Drug: Mitoxantrone Hydrochloride Liposome injection — Mitoxantrone Hydrochloride Liposome injection will be administered by an intravenous infusion on day 1 of each 28-day cycle
  Other Names: Mitoxantrone Hydrochloride Liposome
Drug: Bortezomib for Injection — Bortezomib (1.3 mg/m^2) will be administered by an intravenous injection or subcutaneously on day 1,4,8,11of each 28-day cycle
  Other Names: Bortezomib
Drug: Dexamethasone Acetate Tablets — Dexamethasone (20 mg/d) will be taken orally on day 1,2,4,5,8,9,11,12 of each 28-day cycle
  Other Names: Dexamethasone

SUMMARY:
The purpose of this study is to evaluate the safety and efficacy of mitoxantrone hydrochloride liposome injection in combination with bortezomib and dexamethasone in patients with relapsed or refractory multiple myeloma.

DETAILED DESCRIPTION:
This is a multicenter, open-label, phase I study aimed to evaluate the safety and efficacy of mitoxantrone hydrochloride liposome injection in combination with bortezomib and dexamethasone in patients with relapsed or refractory multiple myeloma. In the study, 60 patients will be recruited into three dose groups. All patients will receive the treatment for the planned 8 cycles(28 days per cycle）until disease progression or unacceptable drug-related adverse events

ELIGIBILITY:
Inclusion Criteria:

1. Patients fully understand and voluntarily participate in this study and sign informed consent;
2. Aged 18-75 years, without gender limitation;
3. Patients with relapsed or refractory multiple myeloma(confirmed by histologically or cytologically) who had received at least one prior line regular treatment;
4. Patients have at least one of the following conditions:（1）Serum M protein≥10g/L;（2）Urine M protein≥200 mg/24h; （3）Serum free light chain(sFLC): κ/λ FLC ratio is abnormal and affected FLC ≥100mg /L
5. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2;
6. Laboratory tests meet the following conditions:

   * Absolute neutrophil count (ANC) ≥1.5x10^9/L (No G-CSF treatment within 1 week prior to the laboratory test);
   * Platelet count ≥ 75x10^9/L (No platelet transfusion within 1 week prior to the laboratory test);
   * Total bilirubin ≤1.5upper limit of normal (ULN);
   * Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 ULN;
   * Creatinine clearance(Ccr) ≥30mL/min.
7. Females of childbearing potential must have a negative serum beta human chorionic gonadotrophin (β-hCG) pregnancy test result prior to enrollment and must agree to use an effective contraception method for the duration of the study treatment and 7 months after the last dose of study therapy.
8. Males patients and their partners must agree to use an effective contraceptive method for the duration of the study treatment and 4 months after the last dose of study therapy.

   -

Exclusion Criteria:

1. Patients with amyloidosis or central nervous system invasion or on dialysis treatment.
2. Life expectancy < 3 months.
3. History of allergy to mitoxantrone hydrochloride or liposomes；or previous treatment with adriamycin or other anthracyclines, with the total cumulative dose (doxorubicin equivalent) ≥350 mg/m^2.
4. History of allergy (except local injection reaction) or intolerance to bortezomib；or one of the following conditions occurred with prior bortezomib regimens: no treatment response (not reach MR)，disease progression within 6 months after the end of last dose.
5. History of contraindications or intolerance to dexamethasone.
6. Any anti-myeloma drug treatment or radiotherapy within 4 weeks prior to the first dose; or enrolled in any other clinical trials of anti-myeloma drug within 3 months prior to the first dose.
7. History of autologous hematopoietic stem cell transplantation within 6 months prior to screening.
8. History of allogeneic hematopoietic stem cell transplantation or solid organ transplantation.
9. Adverse events from the previous treatment have not resolved to ≤ Grade 1 (except for alopecia, hyperpigmentation).
10. Patients with persistent Grade≥2 peripheral neuropathy or Grade 1 peripheral neuropathy with pain.
11. Patients with impaired cardiac function or significant cardiac disease.
12. HBsAg/HBcAb positive with HBV-DNA titer higher than the lower limit of the test value of the research center, or HCV antibody positive with HCV-RNA titer higher than the lower limit of the test value of the research center,or human immunodeficiency virus (HIV) antibody positive.
13. Patients with obvious digestive system dysfunction, which may affect intake, transport and absorption of the study drug.
14. Active bacterial, fungal or viral infections that require systemic treatment within 1 week prior to the first dose
15. Patients underwent major surgery within 6 weeks prior to the first dose, or had a surgical schedule during the study period;
16. History of additional malignant tumor within 5 years, except for locally curable cancer that has been cured.
17. Other medical conditions that, in the judgment of the investigator, may affect the patient's participation in this study.
18. Pregnant or breastfeeding women;
19. Not suitable for this study as decided by the investigator due to other reasons.

    -

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-10-20 (Actual); Primary Completion 2023-04-20 (Estimated); Study Completion 2024-06-20 (Estimated)

PRIMARY OUTCOMES:
Treatment-emergent adverse events (TEAEs) | From the initiation of the first dose to 28 days after the last dose
  To indentify the incidence of TEAEs

SECONDARY OUTCOMES:
Objective response rate (ORR) | Throughout the study treatment(Up to 32 weeks)
  ORR is defined as the proportion of patients who have a best overall response of partial response (PR),very good partial response(VGPR), complete response (CR) or stringent complete response (sCR) as per International Myeloma Working Group (IMWG)
Clinical Benefit Rate(CBR) | Throughout the study treatment(Up to 32 weeks)
  CBR is defined as the proportion of patients who have a best overall response of minimal response(MR),PR,VGPR,CR or sCR as per IMWG
Disease control rate(DCR) | Throughout the study treatment(Up to 32 weeks)
  DCR is defined as the proportion of patients who have a best overall response of stable disease (SD),MR,PR,VGPR,CR or sCR as per IMWG
Duration of response (DoR) | Throughout the study completion.(An average of 12 months)
  DoR is defined as the time from the first assessment of PR,VGPR,CR orsCR until the date of first occurrence of progressive disease (PD) as per IMWG
Progression-free survival (PFS) | Throughout the study completion.(An average of 12 months)
  PFS is defined as the time from the date of first dose until the date of first documented PD as per IMWG or death from any cause, whichever occurs first
Overall survival (OS) | Throughout the study completion.(An average of 36 months)
  OS is defined as the time from the date of first dose until the date of death from any cause

CONTACTS AND LOCATIONS:
Overall Officials: Wenming Chen, Principal Investigator — Beijing Chao Yang Hospital
Locations (1):
- Beijing Chaoyang Hospital, Capital Medical University, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Zhou YL, Zhang JQ, Wang W, Bao L, Fang BJ, Gao D, Su LP, Chen WM, Yang GZ. Bortezomib, Mitoxantrone Hydrochloride Liposome, and Dexamethasone for Relapsed/Refractory Multiple Myeloma: A Multi-Center, Open-Label Phase I Trial. Cancer Med. 2025 Apr;14(8):e70890. doi: 10.1002/cam4.70890. PMID 40232151